CLINICAL TRIAL: NCT00026702
Title: Search for Novel Methods to Detect Acute Renal Failure
Brief Title: Search for New Methods to Detect Acute Renal Failure
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000107; 00-DK-0107
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-30

CONDITIONS: Kidney Disease; Kidney Failure; Kidney Failure, Chronic; Healthy Volunteers; Renal Tubular Toxicity
Keywords: Acute Kidney Injury
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency; Kidney Failure, Chronic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All: Subjects at least three years old

SUMMARY:
The purpose of this study is to find substances in the blood and urine that indicate that a person has kidney damage. It will identify proteins found only in patients with acute kidney failure but not in normal healthy people or in patients with volume depletion.

Adults and children who are at least 3 years old who fall into one of the following four categories may be eligible for this study:

1. Are healthy and have normal kidney function
2. Have volume depletion (this condition differs from acute kidney failure in that it is easily treated with fluids)
3. Are at high risk of kidney failure
4. Have acute kidney failure (kidney shutdown)

All study participants will have a history and physical examination. Up to four blood samples of 3 tablespoons each will be taken for laboratory analysis. Urine will be collected for analysis and to measure urine output. The participants length of stay in the study varies. People with normal kidney function will be in the study for 1 day and patients with volume depletion will be studied 3 days. The length of hospitalization of patients at high risk of kidney failure or in acute kidney failure will depend on the patient s condition and medication requirements.

The results of this study may lead to the development of earlier and more accurate methods for diagnosing acute kidney failure. With earlier detection, treatment could be started earlier, possibly preventing further damage and helping recovery of injury that has already occurred.

...

DETAILED DESCRIPTION:
The mortality of acute renal failure (ARF) remains high despite advances in supportive care. There are no established effective drug therapies, and dialysis may promote renal injury via hypotension or neutrophil activation. Many agents [e.g., mannitol, furosemide, dopamine, Atrial Natriuretic Peptide (ANP), Insulin-like Growth Factor (IGF-1), thyroid hormone, etc.] are effective in animal models but ineffective in treating or preventing human ARF. The failure of these agents in human ARF may be due to late enrollment into the trial; effective therapy will likely require earlier detection.

The objective of this clinical study is to identify new biomarkers of renal injury, progression or recovery by analyzing urinary proteins during ARF. We will enroll patients with ARF, patients at high risk of ARF, patients with volume depletion, patients with urinary tract infection, patients with chronic kidney disease, and normal subjects. The diagnosis of pre-renal versus renal ARF will be made by routine clinical and laboratory testing. The level of renal dysfunction will be determined by creatinine clearance. Those patients at high risk for ARF will be followed prospectively and will undergo additional testing if ARF does develop. Patients will also be studied after creatinine levels return to normal. We will identify protein and/or microRNA biomarkers that are unique to patients with ARF,but not found in normal subjects or patients with volume depletion. It is hoped that some of these proteins may form the basis of new diagnostic tests for ARF.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects >= 3 years old. Both male and female subjects will be recruited without regard to race or ethnic origin.
  2. Either:

     1. Normal (creatinine level < 1.3 mg/dl for adults; creatinine level < standard nomogram for children), OR
     2. Oliguria due to volume depletion (indicated by oliguria and Fractional Excretion of Sodium (FENa) of less than 1%), OR
     3. High risk of ARF, including surgery, transplantation, nephrotoxic antibiotics, or bone marrow transplant. OR
     4. Evidence of ARF as defined by an acute progressive rise in serum creatinine (at least 50% increase within 24 hours preceding enrollment) without stabilization or recovery, despite optimization of hemodynamic fluid status and correction of any known pharmacologic, pre-renal, or post-renal etiologic factors. OR
     5. Urinary tract infection (to serve as control for ARF studies), OR
     6. Established chronic kidney disease (to serve as control for ARF studies).

EXCLUSION CRITERIA:

1. Minors who do not give clear assent, even with parental consent
2. Existence of any other condition which would complicate the implementation or interpretation of the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: subjects with and without kidney disease, can include vulnerable populations such as pregnant women, cognitively impaired adults, or NIH employees
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2000-06-07 (Actual)

PRIMARY OUTCOMES:
estimated GFR | at the time of sample collection
  Serum creatinine will be measured and eGFR will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Star, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-DK-0107.html